CLINICAL TRIAL: NCT04665947
Title: First-in-human Study of the Theranostic Pair [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G in Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Julie L. Sutcliffe, Ph.D, Professor, University of California, Davis
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1667622
Record Dates: First submitted 2020-12-10; First posted 2020-12-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Cancer; Locally Advanced Pancreatic Adenocarcinoma
Keywords: integrin; metastatic pancreatic cancer; PET; theranostic
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a first-in-human 3 + 3 study design to identify dose limiting toxicity and recommended phase 2 dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [177Lu]Lu DOTA-ABM-5G dose escalation therapy study (Experimental): Patients will be undergo [68Ga]Ga DOTA-5G PET/CT scans to confirm eligibility for the [177Lu]Lu DOTA-ABM-5G therapy. Patients with sufficient lesion uptake of [68Ga]Ga DOTA-5G PET/CT will be offered therapy. Escalating doses of 25-200 mCi of [177Lu]Lu DOTA-ABM-5G will be administered in a traditional 3+3 dose escalation design. After escalation, 10 additional patients will be enrolled into a dose expansion cohort.
  Interventions: Drug: [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G.
- Recommended Phase 2 dose [177Lu]Lu DOTA-ABM-5G therapy study (Experimental): Patients will be undergo [68Ga]Ga DOTA-5G PET/CT scans to confirm eligibility for the [177Lu]Lu DOTA-ABM-5G therapy.10 patients will be enrolled in the dose expansion cohort and recieve the highest dose achieved in the [177Lu]Lu DOTA-ABM-5G dose escalation therapy study
  Interventions: Drug: [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G.

INTERVENTIONS:
Drug: [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G. — PET imaging using [68Ga]Ga DOTA-5G will be used to diagnose patients who are eligible for treatment with the [177Lu]Lu DOTA-ABM-5G.
  Other Names: [68Ga]Ga DOTA-5G; [177Lu]Lu DOTA-ABM-5G; [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G theranostic pair

SUMMARY:
This is a Phase I, first-in-human study to evaluate the safety and efficacy of the [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G theranostic pair in patients with locally advanced or metastatic pancreatic adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
This is a Phase I, first-in-human study to evaluate the safety and efficacy of the [68Ga]Ga DOTA-5G /[177Lu]Lu DOTA-ABM-5G theranostic pair in patients with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC). PET imaging using [68Ga]Ga DOTA-5G will be used to diagnose patients who are eligible for the [177Lu]Lu DOTA-ABM-5G. The overall purpose of this study is to identify the dose limiting toxicity (DLT) and recommended phase 2 dose (RP2D) of [177Lu]Lu DOTA-ABM-5G. A 3+3 study design in is proposed to identify the RP2D of [177Lu]Lu DOTA-ABM-5G. An expansion group will receive the RP2D in order to obtain initial estimates of response and additional information on safety of [177Lu]Lu DOTA-ABM-5G.

The hypotheses of this phase I study are that a) [68Ga]Ga DOTA-5G will detect lesions in patients with locally advanced or metastatic pancreas cancer b) the theranostic pair [68Ga]Ga DOTA-5G/ [177Lu]Lu DOTA-ABM-5G will be safe and well tolerated c) we will be able to identify a Recommended Phase 2 Dose (RP2D) for [177Lu]Lu DOTA-ABM-5G therapy to be used in subsequent Phase II trials.

ELIGIBILITY:
Inclusion Criteria:

[68Ga]Ga DOTA-5G PET/CT Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Age 18 or more years
3. Confirmed presence of locally advanced, unresectable or metastatic pancreatic adenocarcinoma (other pancreatic malignant histologies are excluded) with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis)
4. Participant must have documented tumor progression during or following at least one prior systemic regimen as established by CT or MRI scan within 28 days of enrollment
5. Eastern Cooperative Oncology Group Performance Status ≤ 2
6. Participant must have completed prior chemotherapy at least 2 weeks (washout period) prior to [68Ga]Ga DOTA-5G PET scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved to Grade 1 or baseline.
7. Hematologic parameters defined as:

   1. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
   2. Platelet count ≥ 100,000/mm3
   3. Hemoglobin ≥ 8 g/dL
8. Blood chemistry levels defined as:

   1. AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
   2. Total bilirubin ≤ 2 times ULN
   3. Creatinine ≤ 2 times ULN
9. Anticipated life expectancy ≥ 3 months
10. Able to remain motionless for up to 30-60 minutes per scan

[177Lu]Lu DOTA-ABM-5G therapy Inclusion Criteria:

1. Completion of entry into [68Ga]Ga DOTA-5G PET study and completion of scan
2. The presence of at least one measurable disease by [68Ga]Ga DOTA-5G PET/CT (SUVmax>2-fold above normal lung or liver)

Exclusion Criteria:

* [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G therapy Exclusion Criteria:

  1. Participant on any chemical anticoagulant including antiplatelet agents (excluding ASA)
  2. Participants with Class 3 or 4 NYHA Congestive Heart Failure
  3. Clinically significant bleeding within two weeks prior to trial entry (e.g. gastrointestinal bleeding, intracranial bleeding)
  4. Pregnant or lactating women
  5. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days prior to study day 1 or anticipated surgery within the subsequent 6 weeks
  6. Has an additional active malignancy requiring therapy within the past 2 years
  7. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
  8. Psychiatric illness/social situations that would interfere with compliance with study requirements
  9. Previous radiation therapy for the treatment of advanced or metastatic disease
  10. Cannot undergo PET/CT scanning because of weight limits (350 lbs)
  11. INR>1.2; PTT>5 seconds above UNL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
[68Ga]Ga DOTA-5G PET/CT imaging | 2 hours from time of injection
  Assessment of [68Ga]Ga DOTA-5G PET/CT imaging to detect lesions in patients with locally advanced or metastatic pancreatic cancer
[177Lu]Lu DOTA-ABM-5G dose escalation therapy | 30 days from time of injection
  Frequency of dose-limiting toxicities (DLT) of [177Lu]Lu DOTA-ABM-5G at escalating dose levels of [177Lu]Lu DOTA-ABM-5G

SECONDARY OUTCOMES:
Assessment of organ dosimetry of [177Lu]Lu DOTA-ABM-5G | 7-14 days from time of injection
  Assessment of organ dosimetry of [177Lu]Lu DOTA-ABM-5G using SPECT/CT imaging at various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Sutcliffe, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No